CLINICAL TRIAL: NCT05258877
Title: A Single-centre, Open-label, Exploratory Study to Investigate the Pharmacokinetics of Ethionamide and Ethionamide Sulfoxide in Patients Established on Treatment for Tuberculosis.
Brief Title: Pharmacokinetics of Ethionamide and Ethionamide Sulfoxide in Patients Established on Treatment for Tuberculosis.
Status: Completed | Type: Observational
Sponsor: BioVersys AG (Industry)
Collaborators: TASK Applied Science (Other)
Responsible Party: Sponsor
Other Study IDs: Eto-001
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2022-09

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Plasma samples — Up to 80ml of plasma may be collected from each participant over the 24 hour sampling period to be used for PK analysis.

SUMMARY:
To determine the pharmacokinetics of ethionamide (Eto) and ethionamide-sulfoxide (Eto-SO) in participants with tuberculosis (TB) when Eto is dosed under programmatic conditions.

DETAILED DESCRIPTION:
A single-centre, open-label, exploratory pharmacokinetic study. This study is designed to collect blood samples from participants established on a TB treatment regimen which includes Eto. These samples will be analysed for concentrations of Eto and its metabolite Eto-SO.

The medication will not be provided by the study, participants will receive their standard of care medication from their local clinic. Participants will continue to take their total daily dose of Eto on study as prescribed by their primary caregiver, this will not change for their participation on study.

ELIGIBILITY:
Inclusion Criteria:

* Provide written, informed consent prior to all trial-related procedures.
* Male or female, aged between 18 and 65 years, inclusive.
* Receiving Eto as a component of a treatment regimen for tuberculosis for at least one month at the time of enrolment.
* Ability and willingness of participant or legally authorized representative to provide informed consent.

Exclusion Criteria:

* Evidence of clinically significant conditions or findings, other than TB, that might compromise safety of the participant or the interpretation of trial endpoints, per discretion of the Investigator.
* Receiving prohibited concomitant medications (see Prior and Concomitant Medications)
* Evidence of illicit substance use (cannabis, methamphetamines, opiates)
* Pregnant or breastfeeding or planning to become pregnant during the study period.
* Laboratory values: participants with the following laboratory values at screening
* creatinine >1.5 times upper limit of normal [ULN];
* haemoglobin <8.5 g/dL;
* Alanine aminotransferase (ALT) ≥2.0 x ULN;

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pulmonary Tuberculosis
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
To determine the Cmax of ethionamide in participants with tuberculosis (TB) when ethionamide is dosed under programmatic conditions. | 2 days
  maximum observed plasma drug concentration (Cmax)
To determine the Cmax of ethionamide-sulfoxide in participants with tuberculosis (TB) when ethionamide is dosed under programmatic conditions. | 2 days
  maximum observed plasma drug concentration (Cmax)
To determine the AUC of ethionamide in participants with tuberculosis (TB) when ethionamide is dosed under programmatic conditions. | 2 days
  area under the plasma drug concentration versus time (AUC0-24)
To determine the AUC of ethionamide-sulfoxide in participants with tuberculosis (TB) when ethionamide is dosed under programmatic conditions. | 2 days
  area under the plasma drug concentration versus time (AUC0-24)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Dale, Study Chair — BioVersys AG
Locations (1):
- TASK Applied Sciences, Cape Town, South Africa